CLINICAL TRIAL: NCT05043324
Title: Prevention and Treatment of Patient Before, During, and After Covid-19 Infection
Acronym: AntiCov-220
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nguyen Thi Trieu, MD (Individual)
Responsible Party: Sponsor-Investigator, Nguyen Thi Trieu, MD, CEO, Trieu, Nguyen Thi, M.D.
Organization: Trieu, Nguyen Thi, M.D. (Individual)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COVID-19 and Immunodeficiency
Record Dates: First submitted 2021-09-08; First posted 2021-09-14 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Covid19
Keywords: AIDS; HIV; HBV; HCV; Stroke; Metabolic dissorder; Stress
MeSH Terms: conditions — COVID-19; Acquired Immunodeficiency Syndrome; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AntiCov-220 (Experimental): Experimental benefits in resistance to SARS-COV-2 were observed in all patients who had previously received certain components of the AntiCov-220 for various therapeutic purposes.
  Interventions: Drug: AntiCov-220
- AntiCov-220 (Placebo) (Experimental): Experimental benefits in resistance to SARS-COV-2 were observed in all patients who had previously received certain components of the AntiCov-220 (placebo) for various therapeutic purposes.
  Interventions: Drug: AntiCov-220 (placebo)

INTERVENTIONS:
Drug: AntiCov-220 — The daily maintenance, AntiCov-220 dose is to take 3 times a day, 1 tablet each time.
  Other Names: 1a
  Arms: AntiCov-220
Drug: AntiCov-220 (placebo) — The daily maintenance, AntiCov-220 (placebo) dose is to take 3 times a day, 1 tablet each time.
  Other Names: 1b
  Arms: AntiCov-220 (Placebo)

SUMMARY:
AntiCov-220 prevents and treats before, during, and after infection with SARS-CoV-2. The composition is fractionally extracted from herbs (Ascorbic Acid, L-Arginine hydrochloride, Adenosma glutinosum extract, Eclipta prostrata extract, Phyllanthus urinaria extract, Impatiens balsamina extract, Rutin, Pregnenolone acetate, Allium sativum, Pyridoxine 5-phosphate, Cyanocobalamin), using flavonoids, isoflavonoids, and pregnenolone in combination with ascorbic acid as the key compounds in preventing and killing SARS-CoV-2; increase antibodies and protect cells; supplementing precursors to help the body strengthen antibodies and reduce the risk of infection; destroy spike protein, toxic protein, help prevent blood clots causing stroke; restore the physiological function of cells after virus infection; helps the body to stabilize the amount of cortisol in the blood as well as stabilize the production of specific antibodies. The composition participates in anti-inflammatory and cell-protecting processes, bringing blood cortisol, B-lymphocytes, Cyfra 21-1, WBC, CRP, fever, dyspnea, and other signs of respiratory tract inflammation to a normal state and normal limit.

DETAILED DESCRIPTION:
AntiCov-220 can eliminate COVID-19 and its variants at a very early stage when they have not had enough time to multiply and cause disease. AntiCov-220 contains precursors, flavonoids, and special enzymes responsible for protecting human cell membranes and destroying cell membranes of some viruses, especially, COVID-19 cannot replicate in the presence of AntiCov-220 in the body.

AntiCov-220 contains precursors of cortisol. As the investigators know, cortisol has a cell anti-inflammatory, blood pressure regulation, blood sugar regulation, energy booster, and anti-stress roles. It provides precursors to help direct and balance the amount of cortisol in the body that has been imbalanced before.

AntiCov-220 contains flavonoids and Isoflavonoids that are cytoprotective antioxidants, clinically proven to destroy SARS-CoV-2, HBV, HIV, HCV, viruses, reduce complications after COVID-19 infection, prevent neurological sequelae, stroke, cardiovascular sequelae, respiratory sequelae, ...

The anti-inflammatory, stress-reducing, cell-protective, anti-viral, and immunosuppressive processes are performed by an in vivo method that has proven its effectiveness more than ten years ago. AntiCov-220 is an innovative product that can fight against COVID-19 and its variants in the current epidemic situation.

AntiCov-220 is committed to protecting the community of people infected with HBV, HIV, HCV, and SARS-CoV-2 against the risk of the COVID-19 pandemic and its mutations.

AntiCov-220 is easy to implement, highly effective, and helps reduce public health costs, which is essential in protecting human health.

AntiCov-220 can be used alongside current standard treatment regimens prescribed by the World Health Organization.

ELIGIBILITY:
Inclusion Criteria:

* All patients with underlying medical conditions who have been taking medications for these conditions.
* Patients with AIDS, HIV, HBV, HCV, and patients with co-infections.
* The cancer patients are stable.
* Patients with congenital or acquired immunodeficiency.

Exclusion Criteria:

* Unstable cancer patients.

Ages: 16 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Assessment on the level of safety and tolerability of patients against the effects of Covid-19.(Arm 1) | - 18 months
  COVID-19 is a contagious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), Anticov-220 characterized by the targeting and destruction of COVID-19
  * One case of Covid-19 infection with no severe change in a patient with HBeAg (+).
  * A case of HIV/AIDS turns back to HIV. Of the 35 follow-up subjects in this group, 20 were vaccinated and 15 were not. (The two cases mentioned above have not been vaccinated).

SECONDARY OUTCOMES:
Assessment on the level of safety and tolerability of patients against the effects of Covid-19.(Arm 2) | - 18 months
  COVID-19 is a contagious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), Anticov-220 characterized by the targeting and destruction of COVID-19
  _ No one has been infected with Covid-19. Of the 47 follow-up subjects in this group, 40 were vaccinated and 7 were unvaccinated.

CONTACTS AND LOCATIONS:
Overall Officials: Tran Minh Cam Tu, Dr., Principal Investigator — Saigon Biopharma Company Limited
Locations (2):
- Saigon Biopharma LLC, Wilmington, Delaware, United States
- Saigon Biopharma Company Limited, Ho Chi Minh City, Vietnam